CLINICAL TRIAL: NCT00156195
Title: A Phase 3, 12-Month, Extension Study to Evaluate the Safety of Asoprisnil in Subjects With Uterine Leiomyomata
Brief Title: Study to Evaluate the Safety of Asoprisnil in the Treatment of Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M01-391
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Leiomyoma; Menorrhagia; Metrorrhagia
Keywords: Symptomatic Uterine Fibroids; Excessive Uterine Bleeding; Uterine Hemorrhage; asoprisnil
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Hemorrhage | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil

INTERVENTIONS:
Drug: Asoprisnil — 10 mg Tablet, oral Daily for 12 months
  Arms: 1
Drug: Asoprisnil — 25 mg Tablet, oral Daily for 12 months
  Arms: 2

SUMMARY:
The objective of this study is to determine the long-term safety of asoprisnil in women with abnormal uterine bleeding associated with uterine fibroids.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of abnormal uterine bleeding associated with uterine fibroids in women and many women must resort to surgery for relief. The objective of this study is to determine the long-term safety of asoprisnil 10 and 25 mg tablets administered daily for 12 months to women with abnormal uterine bleeding associated with uterine fibroids after an initial 12 months in M01-390 or M01-394. The safety endpoints for this study will be based on assessments of the endometrium, ovarian cysts (if applicable), bone and lipid profiles, adverse events, and changes from baseline laboratory values and vital signs.

Some subjects receiving asoprisnil developed endometrial changes. As a result, dosing was prematurely discontinued for all subjects. To ensure safety, subjects will remain on study and will undergo scheduled study procedures. In most subjects, endometrial changes reversed after asoprisnil discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Women who have completed 12 months of treatment in study M01-390 or study M01-394 and their Visit 12 procedures, respectively
* Otherwise in good health
* Premenopausal based on Estrogen and FSH levels
* Agrees to use of double barrier method of contraception
* Adequate endometrial biopsy with no significant histological disorder

Exclusion Criteria:

* Any abnormal lab or procedure result(s) the study-doctor considers important
* Significant gynecological disorder such as confirmed endometrial polyp
* Hemoglobin < 8.0 g/dL
* History of a blood-clotting disorder
* Any prior surgical and/or invasive procedure(s) for uterine fibroids that resulted in either a cure or made the symptoms go away.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The percent of subjects who demonstrate a clinically meaningful improvement in bleeding and do not require surgical/invasive intervention. | Month 12

SECONDARY OUTCOMES:
The percent of subjects who demonstrate a clinically meaningful improvement in bleeding and do not require surgical/invasive intervention. | Month 6
Change from baseline in menstrual pictogram bleeding score. | Final Month
Change from baseline in the number of days with bleeding. | Final Month
Change from baseline in hemoglobin concentration. | Final Visit
Percent change from baseline in the volume of the largest fibroid. | Final Visit
Change from baseline in bloating, pelvic pressure, dysmenorrhea and urinary symptoms. | Final Visit
Change from baseline in total symptom severity score and the Uterine Fibroid Symptom-Quality of Life total score. | Final Visit
Cumulative percent of subjects who achieve amenorrhea. | Each Month

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott

REFERENCES:
- [Derived] Diamond MP, Stewart EA, Williams ARW, Carr BR, Myers ER, Feldman RA, Elger W, Mattia-Goldberg C, Schwefel BM, Chwalisz K. A 12-month extension study to evaluate the safety and efficacy of asoprisnil in women with heavy menstrual bleeding and uterine fibroids. Hum Reprod Open. 2019 Nov 4;2019(4):hoz027. doi: 10.1093/hropen/hoz027. eCollection 2019. PMID 31777761